CLINICAL TRIAL: NCT01012076
Title: Promoting Development in Toddlers With Communication Delays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Autism Speaks (Other)
Responsible Party: Autism Speaks, Autism Speaks
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G07-02-055-03
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Autism Spectrum Disorder
Keywords: maternal synchrony; parent-child; parent child play; social communication
MeSH Terms: conditions — Autism Spectrum Disorder; Communication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Control (Active Comparator): The active control involves three 90 minute in-home training sessions. These training sessions will be administered by trained graduate students or a postdoctoral student in a developmental psychology or related field. The active control will follow a standardized treatment manual (Kasari, 2008). This treatment manual was based upon the teacher training workshops created by the Center on the Social and Emotional Foundations for Early Learning. Over the course of the intervention, parent and interventionist cover a hierarchy of intervention topics, aiming to improve the parent's ability to successfully promote the child's social and emotional competency.
  Interventions: Behavioral: Active Control vs Experimental Treatment
- Experimental Treatment (Experimental): The parent education program involves 12 in-home training sessions (90 minutes each), is administered by trained graduate and postdoctoral students in developmental psychology or a related field, and follows a standardized treatment manual (Siller, 2005). Over the course of the intervention, parent and interventionist cover a hierarchy of intervention topics, aiming to promote the ability of the parent-child dyad to successfully manage shared toy play.
  Interventions: Behavioral: Active Control vs Experimental Treatment

INTERVENTIONS:
Behavioral: Active Control vs Experimental Treatment — The parent education program involves 12 in-home training sessions (90 minutes each), is administered by trained graduate and postdoctoral students in developmental psychology or a related field, and follows a standardized treatment manual (Siller, 2005). The active control involves three 90 minute in-home training sessions. These training sessions will be administered by trained graduate students or a postdoctoral student in a developmental psychology or related field. The active control will follow a standardized treatment manual (Kasari, 2008). This treatment manual was based upon the teacher training workshops created by the Center on the Social and Emotional Foundations for Early Learning.

SUMMARY:
Eighty parent-child dyads will be recruited and randomly assigned to either the experimental intervention or an active control condition. Subjects assigned to the experimental group will participate in 12 home-based intervention sessions.

DETAILED DESCRIPTION:
The experimental intervention is manualized, follows an illustrated workbook for parents, and uses individualized video-feedback, modeling, and coaching strategies to help parents establish play interactions that promote communication. All participants take part in comprehensive baseline and post-intervention/post-active control assessments, as well as 6- and 12-month follow up assessments. Families in the active control group will also be invited to participate in an oral feedback session to discuss the results from these assessments. Children's involvement in other forms of intervention will be monitored using a validated intervention log so that the moderating effects of these treatments can be examined.

By targeting parent-child interactions, the current intervention ensures that new child behaviors generalize beyond the immediate context of the intervention and are maintained over time (Schreibman, 2000). In addition, by involving parents in the treatment of their children (e.g., by establishing a daily playtime routine), the current intervention ensures that the intervention strategies are implemented with sufficient intensity for causing developmental change (National Research Council, 2001).

ELIGIBILITY:
Inclusion Criteria:

* The child is between 15 and 30 months of age;
* The child scores at least one standard deviation below average on the Social Composite Score of the CSBS DP.

Exclusion Criteria:

* The child has been diagnosed with a known medical condition that has been linked to either autism or mental retardation (e.g., Fragile X, Tuberous Sclerosis, Cerebral Palsy, Hydrocephalus).
* The child has a severe visual, hearing, or motor impairment or fragile health condition that would prevent him/her from validly participating in the assessment procedures.

Ages: 15 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2007-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Maternal Synchronization | 3 months
  Maternal Synchronization will be measured at exit of study.
Maternal Synchronization | 6 months
  Maternal Synchronization will be measured at 6 month follow up of study.
Maternal Synchronization | 12 months
  Maternal Synchronization will be measured at 12 month follow up of study.

SECONDARY OUTCOMES:
Early Social Communication Scale | 3 months
  Early Social Communication Scale will be used to measure joint attention behaviors at exit of study.
Early Social Communication Scale | 6 months
  Early Social Communication Scale will be used to measure joint attention at 6 month follow up.
Early Social Communication Scale | 12 months
  Early Social Communication Scale will be used to measure joint attention at 12 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Connie Kasari, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Hunter College, New York, New York

REFERENCES:
- [Background] Siller M, Sigman M. The behaviors of parents of children with autism predict the subsequent development of their children's communication. J Autism Dev Disord. 2002 Apr;32(2):77-89. doi: 10.1023/a:1014884404276. PMID 12058846
- [Background] Tomasello M, Carpenter M, Call J, Behne T, Moll H. Understanding and sharing intentions: the origins of cultural cognition. Behav Brain Sci. 2005 Oct;28(5):675-91; discussion 691-735. doi: 10.1017/S0140525X05000129. PMID 16262930
- [Background] Siller M, Sigman M. Modeling longitudinal change in the language abilities of children with autism: parent behaviors and child characteristics as predictors of change. Dev Psychol. 2008 Nov;44(6):1691-704. doi: 10.1037/a0013771. PMID 18999331
- [Derived] Kasari C, Siller M, Huynh LN, Shih W, Swanson M, Hellemann GS, Sugar CA. Randomized controlled trial of parental responsiveness intervention for toddlers at high risk for autism. Infant Behav Dev. 2014 Nov;37(4):711-21. doi: 10.1016/j.infbeh.2014.08.007. Epub 2014 Sep 26. PMID 25260191